CLINICAL TRIAL: NCT01189422
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Subcutaneously Administered Teplizumab (MGA031) in Adults With Type 1 Diabetes Mellitus
Brief Title: Subcutaneous Administration of Teplizumab in Adults With Type 1 Diabetes
Acronym: SUBCUE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CP-MGA031-06
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Segment 1: 3 Arms (Experimental)
  Interventions: Drug: teplizumab or placebo
- Segment 2: 4 Arms (Experimental)
  Interventions: Drug: teplizumab or placebo

INTERVENTIONS:
Drug: teplizumab or placebo — infusion or injection

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of subcutaneously administered teplizumab in adults with relatively recent onset T1DM, greater than 12 weeks and less than 52 weeks of presentation of first signs and symptoms of disease to a physician prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Randomization after 12 weeks but within 12 months from first doctor visit for symptoms or signs of diabetes
* Diagnosis of type 1 diabetes mellitus
* Currently receiving insulin therapy
* Detectable fasting or stimulated C-peptide level at screening
* One positive autoantibody test result at screening: Islet-cell autoantibodies (ICA512)/islet antigen-2 (IA-2),Glutamic acid decarboxylase (GAD) autoantibodies, or Insulin autoantibodies

Exclusion Criteria:

* Any medical condition that, in the opinion of the investigator, would interfere with safe completion of the trial
* Previous treatment with monoclonal antibody
* Current treatment with oral antidiabetic agents
* Evidence of active infection

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Dose regimen | 91 days
  Define and evaluate dose regimen based on AEs, PD response and drug levels.